CLINICAL TRIAL: NCT00984958
Title: Bulkamid Treatment of Stress Incontinence in Women With Urinary Stress Incontinence and Not Suitable to TVT-procedure Because of Suspected ISD: A Prospective Randomized Study
Brief Title: Bulkamid Treatment of Stress Incontinence in Women With Urinary Stress Incontinence and Not Suitable to TVT-procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, professor, Skaraborg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bulkamid ISD2009 04
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Urinary Stress Incontinence; Treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Group 1 will get treatment and Group 2 will have no treatment for 2 month
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bulkamid (Other): Injection with Bulkamid
  Interventions: Device: Bulkamid
- expectance (Other): The expectance arm will after 2 month have the same treatment as the treatment arm
  Interventions: Device: Bulkamid expectation

INTERVENTIONS:
Device: Bulkamid — injection of Bulkamid in the urethra
  Arms: Bulkamid
Device: Bulkamid expectation — expectance
  Other Names: after 2 month the patient can be treated
  Arms: expectance

SUMMARY:
The aim of this prospective, randomized study of Bulkamid treatment is to investigate the efficacy of Bulkamid treatment in women with urinary stress incontinence not suitable to TVT-procedure because of suspected ISD.

DETAILED DESCRIPTION:
The aim of this prospective, randomized study is to investigate the effect of Bulkamid injection for women with urinary stress incontinence and not suitable to TVT-procedure because of suspected ISD and compare this treatment with no or traditional treatment. The primary endpoint for efficacy will be reduction of leakage during pad-test at 2 months compared with pad- test before injection.

Secondary endpoints will be patient satisfaction measured at both 2 and 12 months using a questionnaire and the number of side effects.

ELIGIBILITY:
Inclusion Criteria:

Ability to understand the information and to give informed consent.

* At least 50 years of age
* History of urinary leakage during low grade physical activity. A woman with genuine stress incontinence has urinary incontinence during running or jumping. Women with suspected ISD have incontinence at much lower grade of physical activity such as slow walking or standing up and just coughing. Walking, standing up from a chair, and coughing are regarded as low grade of physical activity.
* A positive pad-test (after coughing 10 times) with increase of minimum of 10 grams of urine with 300 ml in the bladder or a 24 h pad-test of more than 100 mg of urine
* No hypermobility of the urethra during cough test.
* Low pressure of the urethra (optional?)
* With a of average miction volume of minimum 150 ml and at least one volume of more than 250

Exclusion Criteria:

* Women with hypermobility of the urethra during coughing and positive Bonney's test
* Women suitable for a TVT procedure.
* Positive urinary culture
* Urge incontinence

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
After 2 months a scheduled visit with a new pad-test will be performed and the questionnaires UDI-6 (lover urinary tract symptoms) and IIQ-7 (quality of life) will be filled in. | 2 month
  less intcontines

SECONDARY OUTCOMES:
After 12 months a scheduled visit with new pad-test will be performed and the questionnaires UDI-6 (lover urinary tract symptoms) and IIQ-7 (quality of life) will be filled in. | 12 month
  less inkontinens

CONTACTS AND LOCATIONS:
Overall Officials: P-G Larsson, professor, Principal Investigator — Departm Ob/Gyn Kärnsjukhuset, 541 85 SKövde, Sweden
Locations (1):
- Deprtm Ob/Gyn, Skövde, Sweden